CLINICAL TRIAL: NCT03691571
Title: Utility of Esophageal Cooling Therapy for the Prevention of Thermal Injury During Atrial Fibrillation Ablation (eCoolAF)
Brief Title: Esophageal Cooling for AF Ablation
Acronym: eCoolAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Attune Medical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 831401
Record Dates: First submitted 2018-09-07; First posted 2018-10-01 (Actual); Results first posted 2021-12-21 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Randomized, blinded single center pilot study
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Esophageal Cooling (Experimental): Patients randomized to Group A receive the EnsoETM (Attune Medical Esophageal Heat Transfer Device).
  Interventions: Device: Esophageal Cooling
- Control (Active Comparator): Patients randomized to Group B receive standard of care treatment (standard temperature probe monitoring).
  Interventions: Device: Control

INTERVENTIONS:
Device: Esophageal Cooling — The EnsoETM is a non-sterile multi-lumen silicone tube placed in the esophagus for the purpose of cooling or warming a patient while simultaneously allowing gastric decompression and drainage.
  Other Names: Attune Medical Esophageal Heat Transfer Device; EnsoETM
  Arms: Esophageal Cooling
Device: Control — Standard of care involves standard temperature probe monitoring.
  Other Names: Standard of care
  Arms: Control

SUMMARY:
The purpose of this study is to determine if esophageal cooling using the Attune Medical Esophageal Heat Transfer Device (EnsoETM) limits the number or seriousness of injury to the esophagus during atrial fibrillation ablation procedures. The EnsoETM is an FDA cleared device used for temperature management, but is not routinely used during atrial fibrillation ablation procedures.

DETAILED DESCRIPTION:
The EnsoETM is a non-sterile multi-lumen silicone tube placed in the esophagus for the purpose of cooling or warming a patient while simultaneously allowing gastric decompression and drainage. Modulation and control of the patient's temperature is achieved by connecting the EnsoETM to an external heat exchanger. Two lumens connect to the external heat exchanger, while a third central lumen provides stomach access for connection to a fluid collection device with low intermittent suction for gastric decompression. The EnsoETM is made of standard medical-grade silicone. It is a single-use, disposable, non-implantable device with an intended duration of use of 72 hours or less. Distilled water circulates within the EnsoETM just like a water blanket.

ELIGIBILITY:
Inclusion Criteria:

1. Patients above the age of 18 years old.
2. Patients with the diagnosis of atrial fibrillation undergoing clinically indicated de-novo AF ablation procedure.
3. Patients must be able to understand and critically review the informed consent form.

Exclusion Criteria:

1. Patients whom are unable to provide informed consent.
2. Patients with contraindication to EGD.
3. History of prior AF ablation procedures.
4. Significant co-morbidities that preclude standard ablation procedure.
5. Patient is ineligible for EnsoETM placement due to:

   * Known esophageal deformity or evidence of esophageal trauma (for example history of esophagectomy, previous swallowing disorders, achalasia).
   * Known ingestion of acidic or caustic poisons within the prior 24 hours.
   * Patients with <40 kg of body mass.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2021-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania - Perelman Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This prospective, randomized, single-center study included patients with symptomatic atrial fibrillation (AF) undergoing first-time radiofrequency catheter ablation between October 2018 and March 2020 at the Hospital of Pennsylvania. Patients were randomized in a 1:1 fashion to achieve esophageal cooling with no luminal esophageal temperature (LET) monitoring (device group) or standard LET monitoring (control group).
Pre-assignment Details: Of 55 enrolled patients, 11 patients withdrew from the study prior to completing the post-procedure endocervical glandular dysplasia (EGD) due to delays obtaining the EGD prior to discharge.
Period: Overall Study
Arm/Group | Esophageal Cooling | Control
Started | 31 | 24
Completed (Eleven patients withdrew from the study prior to completing the post-procedure EGD due to delays obtaining the EGD prior to discharge.) | 22 | 22
Not Completed | 9 | 2
Not completed — Withdrawal by Subject | 9 | 2

BASELINE CHARACTERISTICS:
Population: Fifty-five patients were enrolled in the study with 31 patients randomized to the device group and 24 patients randomized to the control group. Eleven patients withdrew from the study prior to completing the post-procedure EGD due to delays obtaining the EGD prior to discharge and 44 patients completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Esophageal Cooling | Control | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (9.6) | 63.6 (9.3) | 63.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 14 | 16 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.5 (7.3) | 31.0 (5.1) | 30.8 (6.3)
Paroxysmal AF, n (%) [Count of Participants; unit: Participants] | 11 | 14 | 25
LVEF (%) [Mean (Standard Deviation); unit: percentage] | 54.7 (11.4) | 55.8 (9.4) | 55.2 (10.4)
CHA2DS2-VASc Score [Mean (Standard Deviation); unit: risk stratification score 1-9] — Congestive heart failure, hypertension, age ≥75 years, diabetes, stroke, vascular disease, age 65-74, sex class (CHA2DS2-VASc). Calculates stroke risk for patients with atrial fibrillation. Score of 0 is "low" risk of stroke, 1 is "moderate", and any score above 1 is a "high" risk. The CHA2DS2-VASc system, with having three more potential variables, inevitably classifies more patients into a high-risk group.
  risk stratification score 1-9 | 2.2 (1.4) | 2.2 (1.6) | 2.2 (1.5)
Hypertension, n (%) [Count of Participants; unit: Participants] | 12 | 13 | 25
CAD, n (%) [Count of Participants; unit: Participants] | 1 | 4 | 5
Diabetes, n (%) [Count of Participants; unit: Participants] | 1 | 2 | 3
Prior stroke/TIA n (%) [Count of Participants; unit: Participants] | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Participants With Esophageal Thermal Injury
Description: Any injury, occurrence rate measured by EGD
Time Frame: Day 1 to 2
Measure: Count of Participants; unit: Participants
Groups:
- Total: Total number of participants with esophageal thermal injury
Arm/Group | Esophageal Cooling | Control | Total
Number analyzed (Participants) | 22 | 22 | 44
Participants | 8 | 5 | 13
Statistical Analysis 1: Comparison: Total; Esophageal thermal injury was detected in 13/44 (30%) patients; Test type: Superiority; p > .05, Fisher Exact

2. Primary Outcome: Number and Percentage of Participants With Esophageal Injury Based on Severity
Description: The severity of injury measured by EGD
Time Frame: Day 1 to 2
Measure: Count of Participants; unit: Participants
Arm/Group | Esophageal Cooling | Control
Number analyzed (Participants) | 8 | 5
Participants
  Grade 1 - Mild | 1 | 2
  Grade 2 - Moderate | 6 | 0
  Grade 3 - Severe | 1 | 3

3. Secondary Outcome: Posterior Wall Ablation Parameters: Temperature
Description: Catheter Temperature
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: celcius
Arm/Group | Esophageal Cooling | Control
Number analyzed (Participants) | 22 | 22
celcius | 25.0 (1.5) | 25.7 (1.5)
Statistical Analysis 1: Comparison: Esophageal Cooling vs Control; Test type: Other — feasibility/pilot study; p = 0.11, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Posterior Wall Ablation Parameters
Description: Impedance drop (absolute difference)
Time Frame: Day 0
Population: Maximum tissue impedance drop during radiofrequency ablation application as recorded by the electroanatomic mapping system.
Measure: Mean (Standard Deviation); unit: ohms
Arm/Group | Esophageal Cooling | Control
Number analyzed (Participants) | 22 | 22
ohms | 10 (2) | 10 (2)
Statistical Analysis 1: Comparison: Esophageal Cooling vs Control; Test type: Other — feasibility/pilot study; p = 0.73, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Occurrence of Acute PV Reconnection
Description: Number of Participants with Acute PV Reconnection
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | Esophageal Cooling | Control
Number analyzed (Participants) | 22 | 22
Participants | 6 | 1
Statistical Analysis 1: Comparison: Esophageal Cooling vs Control; Test type: Other — feasibility/pilot study; p = 0.10, Fisher Exact

ADVERSE EVENTS:
Time Frame: Approximately 1 month post EGD.
Arm/Group | Esophageal Cooling | Control
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 10/22 | 9/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Esophageal Cooling (N=22) | Control (N=22)
Sore Throat or Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 9
Mild Cough with Trace Blood-Tinged Sputum (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Maximum Core Body Temperature Decrease (Nervous system disorders) | 3 | 0 — The baseline core body temperature in the device group was 36.2±0.8°C and 35.7±1.6°C during active esophageal cooling. The maximum core body temperature decrease observed during active esophageal cool was 0.5±1.2°C.

LIMITATIONS AND CAVEATS:
Pilot study with a relatively small patient pool; Provides an initial assessment regarding the potential clinical benefit of active esophageal cooling for prevention of thermal injury; Fixed ablation parameters and limited to a single ablation catheter technology; Unclear if findings will be reproducible with different ablation strategies or with different ablation technologies. Larger, multi-center studies are needed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/71/NCT03691571/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/71/NCT03691571/ICF_002.pdf